CLINICAL TRIAL: NCT01158547
Title: A Pilot Placebo Controlled, Double-Blind, Randomized Parallel Group Study to Evaluate the Efficacy of Treatment With CLR3001 in Depression
Brief Title: Efficacy Study of CLR3001 in Depression
Status: Completed | Type: Observational
Sponsor: Clera Inc. (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CLR3001
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the ability of CLR3001 to reverse depressive symptoms relatively quickly in adult patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
CLR3001 is thought to work by helping the body's natural responses overcome depression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female out-subjects 18-65 years.
* Single episode or recurrent MDD (to a maximum of 5 prior episodes).
* No current therapy for depression as per washout instructions.
* Able to provide written informed consent.
* Meet criteria for MDD with current MDE through MINI questionnaire.
* Meet criteria for MDD with current MDE, as defined by DSM-IV TR.
* HAMD-17 score ≥ 14 at screening (visit 1) and baseline (Visit 2; Randomization).
* Able to understand and complete questionnaires, and communicate with the investigator and study coordinator.
* Judged to be reliable to keep all appointments and procedures required by the protocol.
* Female subjects of childbearing potential (who are not at least 2 years postmenopausal or surgically sterile or totally abstinent) must be using a reliable, medically acceptable form of contraception and must agree to continue such use throughout the duration of the study. Reliable forms of contraception include oral, implanted, transdermal or injected contraceptives, intrauterine devices, and adequate double barrier methods including use of spermicide. Partner's vasectomy is also an acceptable contraceptive regimen.

Exclusion Criteria:

* Investigators and immediate family members.
* Treatment within the last 90 days with a drug that had not received regulatory approval at the time of study entry.
* Persons who had previously withdrawn from this study or previous study investigating CLR3001.
* A primary diagnosis of Panic Disorder, Social Anxiety Disorder, Obsessive-Compulsive Disorder within the past year.
* The presence of an Axis II disorder, which, in the opinion of the investigator, would interfere with compliance in the study.
* History of active substance dependence within the last half-year, excluding nicotine and coffee, or active substance abuse that may interfere with the outcome of the study.
* Acute suicidal ideation or risk, ≥3 on HAMD-17 suicide item.
* Fall in HAMD-17 score greater than 20% between Visit 1 and Visit 2.
* Serious concomitant diseases such as cancer, serious metabolic (e.g. Insulin dependent diabetes), renal, cardiac, thyroid, immunological, neurological or other significant disease or laboratory abnormality (hematology, blood chemistry, ECG), or treatment for medical conditions which may interact with CLR3001.
* Women who are pregnant or breast-feeding, or men or women who plan to
* Infirmities or living in an area limiting participation in the study or compliance with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2010-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Efficacy using Hamilton Rating Scale for Depression | Weeks 2 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Kennedy, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada